CLINICAL TRIAL: NCT06015763
Title: Correlation Between H.Pylori Colonization and Severity of Gastritis
Brief Title: Correlation Between H.Pylori Colonization and Gastritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Merna Mawgoud Zaki Bechit (Other)
Responsible Party: Sponsor-Investigator, Merna Mawgoud Zaki Bechit, Relation between H.pylori colonization and severity of gastritis, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H.pylori and gastritis
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Gastritis H Pylori
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Endoscopic
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relation between gastritis and H.pylori (Other): Endoscopic
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopic biopsy

SUMMARY:
To study the prevelance rate of H.pylori colonization in patients with gastritis.

To correlate the H.pylori colonization with endoscopic finding. To correlate both H.pylori colonization and endoscopic finding with clinical manifestation.

DETAILED DESCRIPTION:
Helicobacter pylori is a gram negative microaerophilic spiral bacterium that is usually found in the stomach and thereby cause infection , which is associated with varying degrees of damage of superficial and glandular epithelium.

Chronic gastritis is a histological entity that is defined by an inflammatory infiltrate of lymphoblasma cells, cocsometimes polynuclear neutrophils and by progressive glandular atrophy of the gastric mucosa,and probably the main cause of chronic inflammation in the gastric mucosa which is usually caused by H.pylori infection.

In addition to chronic gastritis almost all benign gastroduodenal diseases including peptic ulcer , mucosa associated lymphoid tissue lymphoma and malignant gastroduodenal adenocarcinoma occurs due to previous H.pylori infection that is usually started with gastric precancerous lesion, gastric atrophy , gastric intestinal metaplasia , dysplasia and then turned to gastric carcinoma.

So the evaluation of H.pylori infection status yo non-infection, past infection, current infection by endoscopy has therefore become increasingly important.

The Sydney grading system is one of the most important recognised tools yo charactize histological lesions of chronic gastritis.

The system categorise gastritis according to intensity of mononuclear inflammatory cellular infiltrate , polymorph activity , atrophy , intestinal metaplasia and H.pylori density into mild , moderate and severe categories, but up till now there is non-standard histology reporting formats are still widely used for gastritis and even specialists are often frustrated by the histological definition that make it difficult to identify candidates for clinico-endoscopic surveillance.

Therefore the eradication of this bacterium aimed to interrupt the carcinogenesis process and prevent recurrence of gastritis and peptic ulcer disease.

However despite of the significant researches conducted on H.pylori colonization in gastric mucosa and its association with endoscopic finding and severity of clinical manifestations, and its impact on the Egyptian population is still a topic of debate.

Currently, there is no study has definitively determined this relationship in the Egyptian population despite the high prevalence rate of H.pylori infection

ELIGIBILITY:
Inclusion Criteria:

- All patients with gastritis above 18 years old with chronic H.pylori infection documented by histological examination included in the study.

Exclusion Criteria:

All patients mentioned above who have previous gastrointestinal surgery and patients below 18y .

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between H.pylori colonization and severity of gastritis. | Baseline
  Biopsy will be taken to correlate between severity of gastritis and colonization of H.pylori.